CLINICAL TRIAL: NCT06208124
Title: A Phase 1/2a Study of IMM-6-415 in Participants With Advanced or Metastatic Malignancies Harboring RAS or RAF Oncogenic Mutations
Brief Title: A Study of IMM-6-415 in RAS/RAF Mutant Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Immuneering Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMM6415-101
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumor (Phase 1); Pancreas Adenocarcinoma; Non-small Cell Lung Cancer; Malignant Melanoma (Cutaneous)
Keywords: pan-RAS; pan-RAF; KRAS; NRAS; HRAS; BRAF; targeted therapy; metastatic therapy; RAS; RAF; adenocarcinoma; MEK; dual MEK; G12A; G12C; G12D; G12F; G12V; Q61H; Q61K; Q61R; Q61L; A146T; A146V; K117N; Mitogen-Activated Protein Kinase (MAPK); V600E; V600K
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma, Cutaneous Malignant; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IMM-6-415 (Experimental): Dose Escalation and Dose Expansion
  Interventions: Drug: IMM-6-415

INTERVENTIONS:
Drug: IMM-6-415 — Twice daily, oral tablet administered in 21-day cycles until treatment discontinuation criteria are met.

SUMMARY:
This is a FIH, ascending dose study to characterize the safety, tolerability, optimal dose and preliminary anti-tumor activity of IMM-6-415 in participants with advanced or metastatic solid tumors harboring RAS or RAF oncogenic mutations.

DETAILED DESCRIPTION:
The dose exploration will identify the candidate recommended Phase 2 dose (RP2D) of IMM-6-415 to further explore the anti-tumor activity of IMM-6-415 as monotherapy in Phase 2a tumor-specific cohorts. Patients will be self-administering IMM-6-415 on a daily basis for up to 16 cycles (21-day cycles). During the first 2 cycles, PK and PD will be assessed. Solid tumor types with RAS/RAF mutations are eligible.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Life expectancy >16 weeks
* Part 1: Histologically or cytologically confirmed diagnosis of a locally advanced unresectable or metastatic solid tumor malignancy harboring RAS (NRAS, KRAS, or HRAS)- or RAF- (ARAF, BRAF, RAF1) activating mutations, as documented by genomic analysis. Results of mutation analysis must be available prior to participant enrollment. A prior genomics report from archival tissues or liquid biopsy demonstrating mutation is acceptable
* Part 2: Histologically or cytologically confirmed diagnosis of one of the following locally advanced unresectable or metastatic solid tumor malignancies: pancreatic adenocarcinoma, RASmut melanoma, Class I BRAFmut melanoma, RASmut NSCLC, other RASmut GI cancers (aside from CRC) or any other RAFmut solid tumor as documented by genomic analysis. Results of mutation analysis must be available prior to participant enrollment. A prior genomics report from archival tissues or liquid biopsy demonstrating mutation is acceptable
* Participants must have received at least 1 line of systemic standard-of-care treatment for their advanced or metastatic disease and in the assessment of the Investigator, would be unlikely to tolerate or derive clinically meaningful benefit from other treatment options
* Participants previously treated with codon-specific inhibitors of KRAS (including investigational agents) are eligible
* KRASG12C mutant participants must have received prior treatment with a KRASG12C inhibitor for any approved indication
* Radiologic evidence of measurable disease (i.e., at least 1 target lesion) according to RECIST 1.1 criteria
* ECOG performance status 0 or 1.
* Participant has adequate organ function

Exclusion Criteria:

* Inability to swallow oral medications.
* Symptomatic, untreated, or actively progressing known central nervous system metastases.
* Uncontrolled pleural or pericardial effusion or ascites requiring repeated drainage more than once every 28 days. In dwelling catheters are allowed.
* History of severe COVID-19 infection resulting in current need of supplemental O2 therapy to maintain resting oxygen saturations ≥90%.
* Presence of ongoing toxicities related to prior anticancer therapy that have not resolved to Grade ≤1 and are not otherwise allowed
* Impaired cardiac function or clinically significant cardiac disease
* Uncontrolled intercurrent illness including but not limited to poorly controlled diabetes or any medical condition determined by the Investigator to be a risk
* History or concurrent evidence of retinal vein occlusion (RVO) or current risk factors for RVO. History of clinically significant serous retinopathy, central serous chorioretinopathy or retinal edema.
* History of rhabdomyolysis within 3 months prior to Study Day 1
* HIV-infected participant must be on anti-retroviral therapy and have a well-controlled HIV infection/disease
* Participants with a history of HBV infection no longer requiring treatment are eligible; participants with a history of HCV infection are eligible if HCV viral load is undetectable at screening.
* Females who are pregnant, breastfeeding, or planning to become pregnant and males who plan to father a child while enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Phase 1/2a: Adverse Events | From treatment initiation through 30 days following the last IMM-6-415 dose
  Number of participants with adverse events
Phase 1: Dose-Limiting Toxicities (DLT) | The first 21 days of study treatment
  Number of participants with dose-limiting toxicities
Phase 1: Recommended Phase 2 Dose (RP2D) candidate | Initiation of study treatment through 21 days (up to approximately 18 months)
  Selection of candidate RP2D to take forward into Ph2a
Phase 1: Maximum Observed Plasma Concentration of IMM-6-415 | After 9 weeks (3 Cycles) of study treatment
  Cmax
Phase 1: Time to Reach Maximum Observed Plasma Concentration of IMM-6-415 | After 9 weeks (3 Cycles) of study treatment
  Tmax
Phase 1: Area Under Plasma Concentration (AUC) Time Curve of IMM-6-415 | After 9 weeks (3 Cycles) of study treatment
  AUC0-t
Phase 1: Pharmacodynamic (PD) Activity of IMM-6-415 Plasma Concentrations Over Time | After 9 weeks (3 Cycles) of study treatment
  Surrogate PD Biomarker Assay, pERK
Phase 2a: Overall Response Rate (ORR) | After up to 48 weeks (16 cycles) of study treatment
  The proportion of participants who achieve a best overall response (BOR) of complete response (CR) or partial response (PR), based on RECIST 1.1 criteria

SECONDARY OUTCOMES:
Phase 2a: Maximum Observed Plasma Concentration of IMM-6-415 | After 9 weeks (3 Cycles) of study treatment
  Cmax
Phase 2a: Time to Reach Maximum Observed Plasma Concentration of IMM-6-415 | After 9 weeks (3 Cycles) of study treatment
  Tmax
Phase 2a: Area Under Plasma Concentration (AUC) Time Curve of IMM-6-415 | After 9 weeks (3 Cycles) of study treatment
  AUC0-t
Phase 2a: Disease Control Rate (DCR) | After 12 weeks (4 Cycles) of study treatment
  The proportion of participants who have a best overall response (BOR) of stable disease (SD) or better
Phase 2a: Progression Free Survival (PFS) | Up to approximately 2 years
  The time interval between study treatment start and disease progression or death due to any cause.
Phase 2a: Duration of Response (DOR) | Up to approximately 2 years
  The time interval between an assessment of partial response (PR) or better and disease progression or death due to any cause.
Phase 2a: Landmark 3-Month Survival | After 3 months of study participation.
  The proportion of participants who are still alive after three months on study
Phase 2a: Landmark 6-Month Survival | After 6 months of study participation
  The proportion of participants who are still alive after six months on study
Phase 2a: Overall Survival (OS) | Up to approximately 2 Years
  The time interval between study treatment start and death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Vinny Hayreh, MD, Study Director — Immuneering Corporation
Locations (5):
- United States (5):
  - Honor Health Research Institute, Scottsdale, Arizona
  - City of Hope, Duarte, California
  - Sarah Cannon Research Institute, Denver, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No